CLINICAL TRIAL: NCT02373449
Title: Functional Magnetic Resonance Imaging to Predict and Correlate Clinical Outcomes of Ketamine Infusions for Refractory Neuropathic Pain
Brief Title: Ketamine and fMRI for Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Anuj Bhatia, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-8706-AE
Record Dates: First submitted 2015-02-09; First posted 2015-02-27 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Neuralgia
Keywords: Ketamine; fMRI; refractory neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RS-fMRI (Experimental): All subjects will be instructed to keep their eyes closed but to remain awake during the fMRI measurement. Resting State fMRI (RS-fMRI) will be performed within four weeks of planned infusion of ketamine, immediately after the end of infusion of ketamine on the fifth (last) day of infusion, and on the one month follow-up appointment after the infusion.
  Interventions: Other: RS-fMRI; Drug: Ketamine

INTERVENTIONS:
Other: RS-fMRI — Resting State-functional Magnetic Resonance Imaging. Protocols involving BOLD (blood oxygen level-dependent) and non-BOLD techniques will be used.
Drug: Ketamine — Part of standard care. To be performed over five consecutive days (Monday to Friday) for six hours per day. A therapeutic range of 0.5 to 2.0 mg/kg/hour is targeted.

SUMMARY:
Neuropathic or nerve injury related pain (NP), an extremely unpleasant condition that is difficult to treat, often has a severe, persistent, and unremitting course. Conventional treatments are often ineffective in relieving NP. Recently, the investigators have developed a cost-efficient regimen involving use of low dose infusions of ketamine for treating neuropathic pain in patients in whom oral medications have failed. We have observed excellent benefits in many of these patients. However, this treatment requires titration and monitoring during the infusion and currently it is not possible to predict which patients will benefit from this intervention. The investigators have shown that functional magnetic resonance imaging (fMRI) of the brain can be used as a tool to predict relief of pain and to assess the effect of treatment in some chronic pain conditions. This innovative project involves development of an fMRI-guided treatment with intravenous ketamine in patients with NP. This study aims to analyze patterns of changes in fMRI of the brain, before and after infusion of ketamine and to correlate the changes with pain intensity. The information from this study will help to deliver this therapy earlier to those patients who are most likely to benefit from ketamine.

DETAILED DESCRIPTION:
This trial is exploratory, prospective, non-randomized, single cohort, single-center, with no blinding of participants, treating physicians, and investigators. Study participants undergo a resting-state fMRI before, after and at '1-month post-ketamine infusion' (standard care). Patients will be recruited over 2 years, from Pain Clinics at Toronto Western Hospital and Mount Sinai Hospital. The primary null hypothesis for this trial is that there are no fMRI brain patterns of patients with neuropathic pain that predict pain relief following ketamine infusion. The secondary null hypothesis for this trial is that there are no correlations between specific fMRI brain patterns of patients with neuropathic pain and change in intensity of pain immediately following ketamine infusion. Further secondary hypothesis include that cortical reorganization in the brain as measured by fMRI at one month after the infusion of ketamine does not correlate with persisting analgesic benefit in patients with neuropathic pain. Finally, we hypothesize that ketamine infusions do not provide significant pain relief, reduction in anxiety and depression, and improvement in quality of life early (at 1 month) and late (at 3 months) after the infusions in patients with neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Refractory neuropathic pain diagnosed by a >3 score on DN4 (Douleur Neuropathique 4) questionnaire
* Average daily pain intensity should be moderate or severe, as indicated by a >3 score on NRS (Numerical Rating Scale)
* Duration of neuropathic pain should be more than three months
* Participants should have tried at least three medications for neuropathic pain. Each of these medications should belong to a different pharmacological group: anticonvulsants (gabapentin, pregabalin), tricyclic antidepressants (amitriptyline, nortriptyline, imipramine, desipramine), serotonin noradrenaline reuptake inhibitors (venlafaxine, duloxetine), tramadol, opioids, cannabinoids, methadone, topical lidocaine and capsaicin patches.

Exclusion Criteria:

* Ketamine or lidocaine intravenous infusion within the 6 months preceding enrollment into this trial
* Contraindications to ketamine (allergy, pregnancy, uncontrolled arterial hypertension, uncontrolled hyperthyroidism, severe ischemic heart disease or heart failure, severe liver or kidney disease, space occupying lesion in the brain or the spinal cord, uncontrolled epilepsy and glaucoma)
* Ongoing litigation issues related to the patient's pain that may affect reporting of pain and quality of life
* An unstable medical or psychiatric condition that makes it unsafe to use study medications
* Participants unable to comply with the study protocol (e.g. follow-up visits, filling forms for measuring anxiety, depression, and quality of life)
* Relative (claustrophobia) or absolute contraindications for MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-02; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Correlation between 'baseline (pre-infusion) fMRI patterns' and 'pain relief (>50% pain reduction, as per NRS or 'Numerical Rating Scale')' | 1 month following ketamine infusion

SECONDARY OUTCOMES:
Correlation between 'specific fMRI brain patterns at 1-month post-infusion' and 'change in neuropathic pain intensity (as per NRS) at 3-month post-infusion' | 3 months following ketamine infusion
Change in pain intensity at 1 month post-infusion, as measured by Brief Pain Inventory (BPI) | 1 month following ketamine infusion
Change in pain intensity at 3 months post-infusion, as measured by Brief Pain Inventory (BPI) | 3 months following ketamine infusion
Change in anxiety at 1 month post-infusion, as measured by Hospital Anxiety and Depression Scale (HADS) | 1 month following ketamine infusion
Change in anxiety at 3 months post-infusion, as measured by Hospital Anxiety and Depression Scale (HADS) | 3 months following ketamine infusion
Change in depression at 1 month post-infusion, as measured by Hospital Anxiety and Depression Scale (HADS) | 1 month following ketamine infusion
Change in depression at 3 months post-infusion, as measured by Hospital Anxiety and Depression Scale (HADS) | 3 months following ketamine infusion
Change in quality of life at 1 month post-infusion, as measured by Short Form-36 (SF-36) v2 Health Survey | 1 month following ketamine infusion
Change in quality of life at 3 months post-infusion, as measured by Short Form-36 (SF-36) v2 Health Survey | 3 month following ketamine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, Principal Investigator — UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No